CLINICAL TRIAL: NCT05464160
Title: Focal Muscular Vibration in the Intensive Treatment of Spasticity in Patients with Severe Acquired Brain Injury
Brief Title: Focal Muscular Vibration in Patients with Severe Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, Associated Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4237
Record Dates: First submitted 2022-07-13; First posted 2022-07-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Brain Injuries; Spasticity, Muscle
MeSH Terms: conditions — Brain Injuries; Muscle Spasticity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- G-FMV (Group Focal Muscular Vibration) (Experimental): Patients allocated in the G-FMV, in addition to conventional rehabilitation treatment, will be treated for 3 weeks with FMV, applied to the upper and/or lower limb, depending on the clinical status.
  The G-FMV will perform the treatment at a frequency of 7 times per week for 3 weeks (21 total applications), using the "EVM EVO medical device" (Endomedica, Italy), applying an intensity of 100 Hz for a total of 23 minutes. Specifically, four different trains of stimulation lasting 5 minutes each will be performed, interspersed with 1 minute of rest (20 minutes of treatment + 3 minutes of rest). FMV will be applied on agonist (major spasticity) muscles of the lower limb and/or upper limb, either single-district or multiple-district, according to clinical evidence of intervention. Stimulation will be conducted in a stand-alone session as an adjunctive modality to the rehabilitation project of physiotherapy and occupational therapy.
  Interventions: Device: Focal Muscular Vibration using the EVM EVO medical device (Endomedica, Italy)
- G-CON (Group Conventional) (Active Comparator): Patients allocated in the G-CONwill be treated for 3 weeks by specific conventional rehabilitation based on the clinical status.
  The G-CON will carry out the normal physiotherapy and occupational therapy rehabilitation treatment, as per the rehabilitation project, for an equal total treatment time to the G-FMV. Conventional treatment will focus on joint mobilization, muscle stretching, and neuromuscular facilitation activities, using the main rehabilitation methods (e.g., neurocognitive theory, Bobath Concept, Progressive Neuromuscular Facilitation, etc...)
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Device: Focal Muscular Vibration using the EVM EVO medical device (Endomedica, Italy) — FMV will be applied 7 times per week for 3 weeks (21 total applications), using the "EVM EVO medical device" (Endomedica, Italy), applying an intensity of 100 Hz for a total of 23 minutes.
  Arms: G-FMV (Group Focal Muscular Vibration)
Other: Conventional Rehabilitation — Conventional treatment will focus on joint mobilization, muscle stretching, and neuromuscular facilitation activities, using the main rehabilitation methods (e.g., neurocognitive theory, Bobath Concept, Progressive Neuromuscular Facilitation, etc...)
  Arms: G-CON (Group Conventional)

SUMMARY:
Severe acquired brain injury (sABI) is a group of disorders that cause long-term disability. Rehabilitation is essential to counteract bed immobilization, muscle failure, pain, and sensory deficits that can affect the clinical and rehabilitation pathway of these patients.

Focal muscle vibration (FMV) is a tool that uses low-amplitude, high-frequency vibrations that when applied to muscle-tendon units. This technique, administered at specific frequencies, amplitudes and durations, can generate action potentials of the same frequency as the stimulus applied to the muscle or tendon. This makes it possible to activate selected afferent fibers and stimulate targeted brain areas with persistent effects over time (long-term potentiation).

Regarding the effect of counteracting vibration spasticity, FMV is able to inhibit the reflex arc and induce reciprocal inhibition of functional agonist muscle. In addition, the strong proprioceptive stimulus generated by vibration is able to reach the primary motor and somatosensory cortex, enhancing cortical mechanisms that regulate co-contraction between agonist and antagonist muscles, thereby reducing muscle tone and joint stiffness. In many studies, this technique has been shown to be effective in reducing pain and joint stiffness by improving muscle contraction and motor control.

DETAILED DESCRIPTION:
The present study aims to analyze the effects of focal muscle vibration in patients with sABI. This study is innovative for the setting, as it will take place for the first time within a neurorehabilitation hospital ward, for the intensity of the treatment as patients will undergo daily treatment sessions, for longer periods than protocols so far in the scientific literature. Finally, the cortical effects of the vibratory stimulus will be analyzed through the analysis of cortical neurophysiological correlates

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 years
* Picture of subacute sABI (20 days to 6 months after the acute event), of any etiology (traumatic, vascular, metabolic)
* Presence of spasticity in the affected limb as assessed by the Modified Ashwort Scale (MAS) ≥ 1+

Exclusion Criteria:

* recent treatment with botulinum toxin (within 3 months);
* ongoing treatment with systemic muscle relaxant drugs (baclofen, tizanidine, benzodiazepines);
* deep vein thrombosis;
* central/peripheral accesses ipsilateral to the limb(s) to be treated;
* oncological diseases;
* epilepsy;
* open skin lesions or local infections.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Reduction of spasticity, assessed by Modified Ashworth Scale (MAS) | Change from Baseline MAS at 3 weeks and at 6 weeks
  The Modified Ashworth Scale (MAS) is a scale for the assessment of spasticity consisting of 6 different categories, based on the score assigned in relation to the degree of perceived resistance to passive mobilization.

SECONDARY OUTCOMES:
Reduction of disability, assessed by Disability Rating Scale (DRS) | Change from Baseline DRS at 3 weeks and at 6 weeks
  The Disability Rating Scale (DRS) is a assessment tool through which the degree of disability can be assessed. The DRS consists of 4 categories through which a patient's functional level can be identified. For the category "vigilance and responsiveness" can be scored from 0 to 12, for the category "cognitive skills for self-care" the score ranges from 0 to 9, for the category "dependence on others" from 0 to 5, and for the category "social participation" the score ranges from 0 to 3.
  The total DRS score ranges from 0 (no disability) to 29 (severe vegetative state).
Reduction of disability, assessed by modified Barthel Index (mBI) | Change from Baseline mBI at 3 weeks and at 6 weeks
  The modified Barthel Index (mBI) is a scale used to assess autonomy in activities of daily living.
  It consists of 10 items: "feeding," with a score ranging from 0 to 10; "personal hygiene," with a score ranging from 0 to 5; "bathing or showering," with a score ranging from 0 to 5"; "dressing,",on a score ranging from 0 to 10; "bed/chair transfer," with a score ranging from 0 to 15; "toilet use," with a score ranging from 0 to 10; "bladder," with a score ranging from 0 to 10; "bowel," with a score ranging from 0 to 10; "walking," with a score ranging from 0 to 15; "stairs," with a score ranging from 0 to 10." The mBI score ranges from 0 (fully dependent) to a maximum of 100 (fully dependent).
Reduction of pain, assessed by Faces Pain Scale (FPS) | Change from Baseline FPS at 3 weeks and at 6 weeks
  The FPS is a scale consisting of 11 faces; the faces are represented by an 8 cm × 8 cm black-and-white line drawing. Each face corresponds to a value from 0 (no pain) to 10 (worst possible pain).
Reduction of pain, assessed by Nociception Coma Scale-revised (NCS-r) | Change from Baseline NCS-r at 3 weeks and at 6 weeks
  The Nociception Coma Scale-revised (NCS-r) is an assessment tool developed and validated for measuring nociception and pain in patients with brain injury.
  The NCS consists of four subscales: motor response, verbal response, visual response and facial expression. Each of the subscales is scored from 0 to 3 points, where 3 points equals the maximum possible pain sign for each item. The NCS records the response to noxious stimuli.
Reduction of pain, assessed by Critical-Care Pain Observational Tool (C-POT) | Change from Baseline C-POT at 3 weeks and at 6 weeks
  The C-POT is a nonverbal pain behavior detection tool specifically for ICU patients. It consists of 4 behavioral indicators: facial expression, body movements, respirator adaptation (for intubated patients) or vocalizations (for non-intubated patients), and body tension. Each indicator has three response options (0, 1, or 2), accompanied by a brief description for correct scoring; the total ranges from 0 to 8 (higher scores indicate more intense pain). A total score greater than 3 indicates clinically relevant pain.
Reduction of pain, assessed by Pain Assessment IN Advanced Dementia (Painad) | Change from Baseline Painad at 3 weeks and at 6 weeks
  The Painad is a multidimensional scale of pain assessment, used for patients with marked cognitive impairment or uncooperative. The Painad consists of 5 basic parameters: (i) breathing, (ii) vocalization, (iii) facial expression, (iv) body language, and (v) consolation.
  A score ranging from 0 to 2 is given for each item, in ascending order of observed discomfort. Finally, the sum of the values obtained from each item is performed going to form a score ranging from 0 to 10. A score of 0 indicates no pain; 1 to 3 mild pain; 4 to 6 moderate pain; 7 to 10 severe pain.
Changes in electrocortical activity, assessed by electroencephalogram (EEG) | Change from Baseline EEG at 3 weeks and at 6 weeks
  The information inherent in the assessment of electrocortical activity, using the electroencephalogram (EEG), asking the patient to move the treated limb (or, if not possible, to imagine the movement). The presence of a cortical potential in motor area will be assessed by following the somatotopic organization, by reconstructing a brain map in amplitude;
Changes in muscle activation, assessed by electromyography (EMG) | Change from Baseline EMG at 3 weeks and at 6 weeks
  Through EMG, it is possible to go and record muscle activity

CONTACTS AND LOCATIONS:
Overall Officials: Luca Padua, MD, PhD, Principal Investigator — Fondazione Policlinico Universitaria A. Gemelli IRCCS
Locations (1):
- UOC Neuroriabilitazione ad Alta Intensità, Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alashram AR, Padua E, Romagnoli C, Annino G. Effectiveness of focal muscle vibration on hemiplegic upper extremity spasticity in individuals with stroke: A systematic review. NeuroRehabilitation. 2019 Dec 18;45(4):471-481. doi: 10.3233/NRE-192863. PMID 31868686
- [Background] Lucente G, Valls-Sole J, Murillo N, Rothwell J, Coll J, Davalos A, Kumru H. Noninvasive Brain Stimulation and Noninvasive Peripheral Stimulation for Neglect Syndrome Following Acquired Brain Injury. Neuromodulation. 2020 Apr;23(3):312-323. doi: 10.1111/ner.13062. Epub 2019 Nov 14. PMID 31725939
- [Background] Marconi B, Filippi GM, Koch G, Giacobbe V, Pecchioli C, Versace V, Camerota F, Saraceni VM, Caltagirone C. Long-term effects on cortical excitability and motor recovery induced by repeated muscle vibration in chronic stroke patients. Neurorehabil Neural Repair. 2011 Jan;25(1):48-60. doi: 10.1177/1545968310376757. Epub 2010 Sep 12. PMID 20834043
- [Background] Murillo N, Valls-Sole J, Vidal J, Opisso E, Medina J, Kumru H. Focal vibration in neurorehabilitation. Eur J Phys Rehabil Med. 2014 Apr;50(2):231-42. PMID 24842220
- [Background] Noma T, Matsumoto S, Shimodozono M, Etoh S, Kawahira K. Anti-spastic effects of the direct application of vibratory stimuli to the spastic muscles of hemiplegic limbs in post-stroke patients: a proof-of-principle study. J Rehabil Med. 2012 Apr;44(4):325-30. doi: 10.2340/16501977-0946. PMID 22402727